CLINICAL TRIAL: NCT05229991
Title: Once Daily (QD) Dosing of Lonafarnib (LNF) Co-administered With Ritonavir (RTV) for Treatment of Chronic Hepatitis D Virus Infection
Brief Title: Once Daily Dosing of Lonafarnib Co-administered With Ritonavir for Treatment of Chronic Hepatitis D Virus Infection
Acronym: LOWR6
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Soroka University Medical Center (Other)
Collaborators: Eiger BioPharmaceuticals (Industry)
Responsible Party: Principal Investigator, Ohad Etzion, Director, Department of Gastroenterology & Liver Diseases, Soroka University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SOR-0527-20-CTIL; SCRC20042 (Other: Soroka Clinical Research Center)
Record Dates: First submitted 2022-01-27; First posted 2022-02-08 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Hepatitis D, Chronic
Keywords: Hepatitis D; Lonafarnib; Ritonavir; Hepatitis B
MeSH Terms: conditions — Hepatitis D, Chronic; Hepatitis D; Hepatitis B | interventions — lonafarnib; Ritonavir

STUDY DESIGN:
Intervention Model Description: LNF50/RTV200 QD will be administered orally, over a 48-week treatment period, with a 24-week post-treatment follow-up period, in patients with chronic HDV infection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Lonafarnib 50mg co-administered with ritonavir 200 mg
  Interventions: Drug: Lonafarnib; Drug: Ritonavir

INTERVENTIONS:
Drug: Lonafarnib — once-daily dosing of lonafarnib 50 mg with ritonavir 200 mg over a 48-week treatment period.
  Other Names: LNF
Drug: Ritonavir — once-daily dosing of lonafarnib 50 mg with ritonavir 200 mg over a 48-week treatment period.
  Other Names: Norvir

SUMMARY:
Open label, single arm, multi-center clinical trial of lonafarnib 50 mg QD plus ritonavir 200 mg QD, administered orally, over a 48-week treatment period, with a 24-week post-treatment follow-up period, in patients with chronic Hepatitis D Virusinfection.

Objectives: To evaluate the safety and tolerability of once daily dosing of lonafarnib 50 mg with ritonavir 200 mg over a 48-week treatment period.

To evaluate the effect of once daily dosing of lonafarnib 50 mg with ritonavir 200 mg over a 48-week treatment period with a 24-week post-treatment follow-up on HDV viral levels.

Trial population: Up to 30 patients with chronic HDV infection with detectable HDV RNA and compensated liver disease.

DETAILED DESCRIPTION:
Background: Hepatitis D virus (HDV) was identified as the infectious agent causing viral hepatitis in the presence of hepatitis B virus (HBV). While HDV can replicate autonomously inside the hepatocyte, the virus requires co-infection with HBV to complete virion assembly and to facilitate transmission. HDV causes the most severe form of viral hepatitis, with rapid progression to cirrhosis and high rates of development of hepatocellular carcinoma. Currently there are no FDA approved therapies for chronic HDV infection (CHD) which presents an unmet medical need. The off-label use of pegylated interferon alpha (Alpha) for the treatment of CHD has so far been explored in several small single-arm studies and in 2 randomized controlled clinical trials, showing limited efficacy and high relapse rates. In addition, Alpha is associated with a poor tolerability profile and its use is limited in patients with advanced disease.

Lonafarnib (LNF), a FT inhibitor has been evaluated in over 2,000 subjects in clinical studies, comprising more than fifty Phase 1 and Phase 2 studies and two Phase 3 studies, with healthy subjects and patients with HDV, cancer, Hutchinson-Gilford progeria syndrome (HGPS) and progeroid laminopathies. Treatment with LNF has been administered as continuous (up to 11 years in HGPS) and intermittent therapy (exceeding one year in cancer patients).

The use of LNF in CHD has been assessed in a proof of concept study, a series of four phase 2 clinical trials (the LOWR program) and an on-going phase 3 clinical trial (D-LIVR study).

Hypothesis: that treatment with LNF50/RTV200 QD for 48 weeks will be safe and lead to a reduction in HDV RNA levels at end of treatment and end of follow up.

Procedures: At baseline, systems review, physical examination, vital signs (temperature, blood pressure, pulse rate per minute), anthropometric measurements (weight, height and BMI) and ECG will be performed. Information regarding the use of alcohol and drugs, symptoms and use of concomitant medications collected. Blood will be drawn for testing of local CBC, chemistry, coagulation studies, HDV antibody and RNA levels, HCV antibody (& RNA if necessary), HBsAg levels, HBeAg status, HBV DNA levels, liver elastography and ultrasound. All blood tests besides HDV RNA levels, will be performed at a local lab. HDV RNA level testing will be performed at a central laboratory. Pregnancy test will be performed in females of child-bearing potential. Trial medications will be dispensed. Use of anti-HBV therapy (tenofovir or entecavir) will be confirmed.

Follow up visits will be conducted at week 4, 12, 24, 36 and 48 of treatment and at 24 weeks after stopping treatment and will include systems review, ECG recordings, evaluation of concomitant medications use, adverse events monitoring and assessment of compliance with trial medications and anti HBV therapy. In addition, blood will be drawn for measurement of CBC, chemistry panel, coagulation tests and HDV RNA and HBV DNA levels at each visit. Trial medications will be dispensed at each visit during the treatment phase of trial.

Adverse events and concomitant medications will be collected throughout the trial.

Data to capture:

* Demographic data: Gender, age, ethnicity, country of birth
* Detailed medical history: including currently prescribed medications, recently administered medications, dispensing date, past medications use and dispensing date, past medical diagnosis including diagnosis date, past medical procedures including procedure date, allergies.
* Habits: history of recreational drugs and alcohol consumption (using CAGE questionnaire).
* Clinical evaluation: Systems review, anthropometric measurements (weight, height and BMI), physical examination, vital signs, symptom questionnaire and AE assessment.
* Blood tests: Complete blood count, biochemistry panel, coagulation tests, anti-HDV antibody, anti HCV antibody, HDV RNA, HBV DNA.

Safety data collected during the trial (e.g., AEs and laboratory test results) will be monitored on an ongoing basis by the trial team.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic HDV infection, with compensated liver disease, documented by a positive HDV antibody (Ab) test and HDV RNA by quantitative polymerase chain reaction (qPCR) assay, prior to initiation of trial treatment.
2. Demonstrable suppression of HBV DNA (< 100 IU/mL) following anti-HBV nucleos(t)ide treatment prior to initiating trial therapy.
3. Willing and able to comply with trial procedures and provide written informed consent.
4. ALT > ULN documented on at least one occasion during the 12 months preceding enrollment to the trial.
5. Male and female participants who are 18 years of age or above.
6. ECGs demonstrating no acute ischemia or clinically significant (CS) abnormality and a corrected QT interval by Fridericia correction formula (QTcF) < 450 ms in males and <470 ms in females.
7. Sexually active female patients of childbearing potential and sexually active male patients with partners of childbearing potential must agree to use adequate methods of contraception during the trial. Females of childbearing potential are all those except women who are surgically sterile, who have medically documented ovarian failure, or who are at least 1 year postmenopausal.

For female patients:

* Progestin-based hormonal contraception (implant, injection, oral) associated with inhibition of ovulation for ≥ 3 months before screening. Use of a progestin-based implant or injection method requires the additional use of a barrier method (use of condom [male partner] or diaphragm with spermicide or cervical cap with spermicide) from screening. Use of a progestin-only, oral method requires the additional use of double barrier methods (use of condom [male partner] with either diaphragm with spermicide or cervical cap with spermicide) from screening, or
* Intrauterine device (IUD) or intrauterine system (IUS) in place ≥ 3 months before screening AND a barrier method (use of condom [male partner] or diaphragm with spermicide or cervical cap with spermicide) from screening, or
* Surgical sterilization of the partner (vasectomy ≥ 1 month before screening) AND a barrier method (use of condom [male partner] or diaphragm with spermicide or cervical cap with spermicide) from screening, or
* Double-barrier methods (use of condom [male partner] with either diaphragm with spermicide or cervical cap with spermicide) from screening.

For male patients:

* Surgical sterilization (vasectomy ≥ 1 month before screening) AND a barrier method (use of condom or diaphragm with spermicide or cervical cap with spermicide) from screening, or
* Consistently and correctly use a condom from screening AND female partner must agree to use a hormonal contraceptive, a nonhormonal non-barrier method (eg, copper IUD), or a nonhormonal barrier method (eg, diaphragm with spermicide or cervical cap with spermicide).

Exclusion Criteria:

1. Participation in a clinical trial with, or use of, any investigational agent within 30 days or 5 half-lives, whichever is longer, before starting LNF treatment.
2. Female patients who are pregnant or breastfeeding. Female patients must have a negative serum test at screening and a negative urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [hCG] at baseline, within 24 hours prior to the start of any investigational agent). Male patients with female sexual partners who are pregnant.
3. Current or previous history of decompensated liver disease (e.g. variceal bleeding, ascites, hepatic encephalopathy, hepatorenal syndrome).
4. Platelet count < 70,000 cells/mm3; white blood cell (WBC) < 3,000 cells / mm3
5. Creatinine clearance (< 30 mL/min by Cockroft-Gault).
6. Co-infected with human immunodeficiency virus (HIV) or hepatitis C virus (HCV). Patients with a positive HCV Ab at baseline are allowed if they have completed a curative antiviral regimen and have documented undetectable HCV RNA 12 weeks or more following last dose of anti-HCV medications.
7. Abnormal thyroid-stimulating hormone (TSH) or free thyroxine (fT4) levels. Patients with well-controlled thyroid function or TFTs that are not clinically significant may be enrolled.
8. Evidence of another form of viral hepatitis or another form of liver disease (eg, autoimmune liver disease, primary biliary cirrhosis, primary sclerosing cholangitis, Wilson's disease, alcoholic liver disease, nonalcoholic steatohepatitis, hemochromatosis, alpha 1 anti-trypsin deficiency).
9. History of hepatocellular carcinoma.
10. Retinal disorder or clinically relevant ophthalmic disorder
11. Any malignancy within 5 preceding years. Exceptions are malignancies surgically excised with curative intent and/or evidence of being disease free for at least 5 years (eg, breast ductal carcinoma in situ [DCIS] or squamous/basal cell skin cancer treated with curative intent), or successfully treated in-situ carcinoma of the cervix
12. Other significant medical condition that may require intervention during the trial.
13. Any condition that may impact proper absorption (eg, short bowel syndrome, inflammatory bowel disease, atrophic gastritis, partial gastrectomy) should be discussed with the Medical Monitor.
14. Consumption of grapefruit, Seville oranges, or product that contains grapefruit or Seville oranges.
15. Use of heparin or warfarin during the trial.
16. Long-term treatment (> 2 weeks) before or during the trial with agents that have a high risk for nephrotoxicity or hepatotoxicity.

    1. Concomitant use (within 2 weeks of Day 1 and throughout trial conduct) of any medications (prescription, OTC, herbal products) or foods as follows:
    2. Known potent inhibitors of CYP3A, including statins (with the exception of pravastatin and fluvastatin);
    3. Known potent inducers of CYP3A or CYP3A sensitive substrates;
    4. Known CYP2C19 and P-gp sensitive substrates with a narrow therapeutic index - refer to the Concomitant Medication Manual for additional instructions;
    5. Known sensitive substrates of OCT1 with a narrow therapeutic index; and
    6. Drugs known to prolong the PR or QT interval unless otherwise described in this protocol.
17. Concomitant use of medications contraindicated in the prescribing information for RTV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Viral load change | 48 weeks
  Change from baseline in HDV viral load at end of treatment
Viral load change | 72 weeks
  Change from baseline in HDV viral load at end of follow-up

SECONDARY OUTCOMES:
HDV RNA levels below LLOQ | 72 weeks
  Proportion of patients with HDV RNA levels below limit of quantification (LLOQ) at end of treatment and end of follow up
Viral load change | 24 weeks
  Change from baseline in HDV viral load at weeks 4, 12 and 24

OTHER OUTCOMES:
Safety: Rate of treatment-emergent and treatment-related severe adverse events | 72 weeks
  Number of severe adverse events related to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ohad Etzion, MD, Principal Investigator — Soroka University Medical Center
Locations (3):
- Soroka UMC, Beersheba, Israel
- New Zealand Liver Transplant Unit, Auckland City Hospital, Auckland, New Zealand
- Department of Gastroenterology and Hepatology, Koç University Medical School, Istanbul, Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No